CLINICAL TRIAL: NCT05302973
Title: Effects of Aerobic Exercise in People With Post-COVID-19: a Randomized Controlled Trial
Brief Title: Aerobic Exercise in People With Post-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2592 CE
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: aerobic exercise; rehabilitation; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (Active Comparator): Inpatient rehabilitation - person-centred and tailored to individual participant needs - which take into account the different sequelae associated with the severity of COVID-19, the prolonged stay of people in the acute hospital or in the intensive care unit, and the pre-existing comorbidities.
  Interventions: Other: Conventional rehabilitation
- Aerobic exercise (Active Comparator): Addition of aerobic exercise to conventional inpatient rehabilitation treatment for people wtih post-COVID-19.
  Interventions: Other: Conventional rehabilitation; Other: Aerobic exercise

INTERVENTIONS:
Other: Conventional rehabilitation — 1h/day for 5 days/week of conventional rehabilitation for people wtih post-COVID-19
Other: Aerobic exercise — 30 min/day of aerobic exercise added to 1h/day for 5 days/week of conventional rehabilitation for people wtih post-COVID-19
  Arms: Aerobic exercise

SUMMARY:
The primary aim of this study is to study the feasibility of an aerobic training, in addition to conventional rehabilitation, in patients post sequela of interstitial pneumonia due to COVID-19. In particular, we wish to verify if patients could tolerate this kind of physical activity and if there are any adverse effects. The secondary aim is to evaluate if the aerobic exercise is effective in improving functional capacity and gait performance in these patients respect to the common physiotherapy.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) is an infectious disease caused by SARS-CoV-2 that mainly affects the respiratory system (Landi et al., 2020). While the majority (80%) of people infected with COVID-19 presents mild to moderate disease (Huang et al., 2020; Rodriguez-Morales et al. 2020), for a considerable number of subjects, generally >65 years and with comorbidities, the infection can have very serious sequelae (about 20%) (Yang et al., 2020). Of those requiring hospitalization, a high portion (20%) require management in the intensive care unit (ICU) often for an acute respiratory distress syndrome (ARDS) (Simpson and Robinson, 2020).

People with critical illness due to COVID-19 has not only a disease primarily affecting the lung, but present also a multi-organ involvement (Gemelli Against COVID-19 Post-Acute Care Study Group, 2020). During periods of critical illness and hospitalization, it is common to experience a loss of physical function (Rawal et al., 2017), characterized by the development of new or worsening of existing impairments. This decrease in physical functioning is thought to be attributed to prolonged periods of immobility, during which time people experience deconditioning, develop critical illness, polyneuropathy and myopathy (Rooney et al., 2020). This results in a motor disability and a reduction of independence in the activities of daily living (ADL) (Abate et al., 2020; Rodriguez-Morales et al. 2020; Herridge et al. 2011; Barnato et al., 2011).

Several authors reported that people with COVID-19 - even without motor limitation prior to hospitalization - in the post-acute phase show muscle weakness, reduced physical performance, exercise-induced oxygen desaturation and hampered performance of ADLs still when discharged home (Belli et al., 2020; Paneroni et al., 2020). In those with severe and critical COVID-19 course, the impairments in pulmonary function and physical performance may be identified four months after the infection (Guler et al., 2021). These findings suggest that there is a clear need to plan for post-acute and chronic rehabilitation for people recovering from COVID-19 (Barker-Davies et al., 2020).

People with COVID-19 are heterogeneous, with different manifestations and comorbidities, and show disabling sequelae when recovering from the infection. Consequently, rehabilitation, which is necessary for facilitating the recovery and the discharge to home, has to be patient-centered and tailored to individual patient needs and impairments (Barker-Davies et al., 2020).

Therefore, it may be useful to conduct a prospective longitudinal study on subjects with COVID-19 who have undergone a period of hospitalization for severe or critical COVID-19 and who were discharged from the post-acute ward to a rehabilitation post-COVID-19 ward. Moreover, since experts strongly recommended a low-/moderate-intensity physical exercise in the first weeks following hospitalization in the COVID wards (Spruit et al., 2020), there is the need to consider the addition of an aerobic exercise training to the usual rehabilitation.

The primary purpose of this randomized controlled clinical trial is to verify the experimental aerobic training may be feasible in subjects with a sequela of interstitial pneumonia due to COVID-19 (people with post-COVID-19) and performed without the manifestation of serious adverse events.

The secondary purpose is to verify whether the addition of aerobic activity can increase physical performance compared to a program in which no aerobic activity is foreseen.

ELIGIBILITY:
Inclusion Criteria:

1. Defined diagnosis of interstitial pneumonia due to COVID-19;
2. Two negative nasopharyngeal swab test for SARS-CoV-2;
3. Functional independence before the COVID-19;
4. Mini-mental state examination (MMSE) score > 24.

Exclusion Criteria:

1. Positivity to COVID-19;
2. Patients living in a nursing home or not autonomous prior to the COVID-19;
3. Presence of moderate or severe heart disease (Grade III or IV, New York Heart Association);
4. Presence of neurological disease;
5. Low compliance;
6. Patients with low rehabilitation needs (FIM total score at admission >100)
7. Terminal illness (life expectation <6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Analysis of feasibility | Up to 2 weeks
  To assess the feasibility, it will be evaluated the adherence to treatment of participants enrolled in the aerobic exercise group. It will be expressed both as compliance rates, defined in terms of duration (% sessions performed reaching the goal of 30min) and prescribed intensity (% sessions performed at an intensity between 64-76% HRmax).

SECONDARY OUTCOMES:
Timed Up and Go (TUG) test | Up to 2 weeks
  TUG is a physical functional measure in which subjects are asked to stand up from a chair, walk 3 m to a horizontal line marked with tape on the floor, turn around, walk back and sit down at a comfortable pace (Podsiadlo and Richardson, 1991). Time in seconds necessary for perform the test will be collected.
Muscle torque of knee extensors | Up to 2 weeks
  The muscle torque of the knee extensors will be evaluated pre- and post-training with the use of a handheld dynamometer. The patient will be required to perform a sub-maximal contraction in knee extension, followed by two maximal contractions during which the physiotherapist will give verbal encouragement. The evaluation will be performed first on one limb, then on the other, with a 30-second pause between one contraction and the next. The mean value of the two right- leg and left-leg tests will be recorded. Measurements will be converted from kilo to newton.
Handgrip strength | Up to 2 weeks
  The handgrip strength will be measured bilaterally with a calibrated Jamar dynamometer. In accordance with the recommendations of the American Society of Hand Therapist, subjects will be seated with feet flat on the floor, the tested arm adducted against the body in neutral rotation, the elbow in 90° of flexion, and the forearm in neutral rotation pronation/supination (Fess and Moran, 1981). Two trials for each arm will be performed; the average of the right and left force will be recorded by the tester in kilo and then converted to newtons.
1-minute sit-to-stand test (1STST) | Up to 2 weeks
  The 1STST is a widely implementable measure of lower body muscular strength and endurance (Bohannon, 1995) which capture the number of stands a person can complete in 1 minute without using the arms. Patients will be asked to perform repetitions of standing upright and then sitting down in the same position at a self-paced speed (safe and comfortable) as many times as possible for 1 min, without using the arms and fully sitting between each stand. The number of completed stands will be recorded. SpO2 before and after the test will be recorded.
Cumulated Ambulation Score - Italian version (CAS-I) | Up to 2 weeks
  The CAS-I is a 3-item scale assessing activities that characterize the patient's basic mobility skills: 1) getting in and out of bed, 2) sit-to-stand from a chair with armrests and 3) walking indoors with the use of appropriate walking aids. Each activity is assessed on a three-point ordinal scale from 0-2 (0 = Not able to, despite human assistance and verbal cueing, 1 = Able to, with human assistance and/or verbal cueing from one or more persons, 2 = Able to safely, without human assistance or verbal cueing, use of a walking aid allowed) resulting in a total daily CAS score ranging from zero to six.
Functional Independence Measure (FIM) | Up to 2 weeks
  This scale is a widely used tool for rating the rates patients' ADL performances. It is composed by 18 items, that is 13 motor and 5 cognitive items, each of whom is assigned a score between 7 (total independence) and 0 (total dependence). Therefore, the total FIM scores range between 18 (reflecting complete functional dependency) and 126 (reflecting complete functional independency).
Physical Activity Scale for the Elderly (PASE) | Up to 100 days
  It is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiologic studies of persons age 65 years and older. The PASE score combines information on leisure, household, and occupational activity (Washburn et al., 1993).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Corna, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri SpA
Locations (1):
- Istituti Clinici Scientifici Maugeri, Veruno, Novara, Italy

REFERENCES:
- [Background] Abate SM, Ahmed Ali S, Mantfardo B, Basu B. Rate of Intensive Care Unit admission and outcomes among patients with coronavirus: A systematic review and Meta-analysis. PLoS One. 2020 Jul 10;15(7):e0235653. doi: 10.1371/journal.pone.0235653. eCollection 2020. PMID 32649661
- [Background] Barnato AE, Albert SM, Angus DC, Lave JR, Degenholtz HB. Disability among elderly survivors of mechanical ventilation. Am J Respir Crit Care Med. 2011 Apr 15;183(8):1037-42. doi: 10.1164/rccm.201002-0301OC. Epub 2010 Nov 5. PMID 21057004
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] Belli S, Balbi B, Prince I, Cattaneo D, Masocco F, Zaccaria S, Bertalli L, Cattini F, Lomazzo A, Dal Negro F, Giardini M, Franssen FME, Janssen DJA, Spruit MA. Low physical functioning and impaired performance of activities of daily life in COVID-19 patients who survived hospitalisation. Eur Respir J. 2020 Oct 15;56(4):2002096. doi: 10.1183/13993003.02096-2020. Print 2020 Oct. PMID 32764112
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Fess E, Moran C. Clinical assessment recommendations: American Society of Hand Therapists. Chicago: The Society; 1981.
- [Background] Gemelli Against COVID-19 Post-Acute Care Study Group. Post-COVID-19 global health strategies: the need for an interdisciplinary approach. Aging Clin Exp Res. 2020 Aug;32(8):1613-1620. doi: 10.1007/s40520-020-01616-x. Epub 2020 Jun 11. PMID 32529595
- [Background] Guler SA, Ebner L, Aubry-Beigelman C, Bridevaux PO, Brutsche M, Clarenbach C, Garzoni C, Geiser TK, Lenoir A, Mancinetti M, Naccini B, Ott SR, Piquilloud L, Prella M, Que YA, Soccal PM, von Garnier C, Funke-Chambour M. Pulmonary function and radiological features 4 months after COVID-19: first results from the national prospective observational Swiss COVID-19 lung study. Eur Respir J. 2021 Apr 29;57(4):2003690. doi: 10.1183/13993003.03690-2020. Print 2021 Apr. PMID 33419891
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Landi F, Barillaro C, Bellieni A, Brandi V, Carfi A, D'Angelo M, Fusco D, Landi G, Lo Monaco R, Martone AM, Marzetti E, Pagano F, Pais C, Russo A, Salini S, Tosato M, Tummolo A, Benvenuto F, Bramato G, Catalano L, Ciciarello F, Martis I, Rocchi S, Rota E, Salerno A, Tritto M, Sgadari A, Zuccala G, Bernabei R. The New Challenge of Geriatrics: Saving Frail Older People from the SARS-COV-2 Pandemic Infection. J Nutr Health Aging. 2020;24(5):466-470. doi: 10.1007/s12603-020-1356-x. No abstract available. PMID 32346682
- [Background] Paneroni M, Simonelli C, Saleri M, Bertacchini L, Venturelli M, Troosters T, Ambrosino N, Vitacca M. Muscle Strength and Physical Performance in Patients Without Previous Disabilities Recovering From COVID-19 Pneumonia. Am J Phys Med Rehabil. 2021 Feb 1;100(2):105-109. doi: 10.1097/PHM.0000000000001641. PMID 33181531
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Rawal G, Yadav S, Kumar R. Post-intensive Care Syndrome: an Overview. J Transl Int Med. 2017 Jun 30;5(2):90-92. doi: 10.1515/jtim-2016-0016. eCollection 2017 Jun. PMID 28721340
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Rooney S, Webster A, Paul L. Systematic Review of Changes and Recovery in Physical Function and Fitness After Severe Acute Respiratory Syndrome-Related Coronavirus Infection: Implications for COVID-19 Rehabilitation. Phys Ther. 2020 Sep 28;100(10):1717-1729. doi: 10.1093/ptj/pzaa129. PMID 32737507
- [Background] Simpson R, Robinson L. Rehabilitation After Critical Illness in People With COVID-19 Infection. Am J Phys Med Rehabil. 2020 Jun;99(6):470-474. doi: 10.1097/PHM.0000000000001443. PMID 32282359
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031